CLINICAL TRIAL: NCT05594004
Title: A Meta-analysis Comparing Electric and Manual Toothbrushes on Plaque Removal and Gingival Health
Brief Title: A Meta-analysis Comparing Toothbrushes on Plaque Removal and Gingival Health
Status: Completed | Type: Observational
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022BrushMetaAnalysis
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Gingivitis; Dental Plaque
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oscillating-Rotating electric toothbrush: Twice daily brushing
  Interventions: Device: Oscillating-rotating electric toothbrush
- Sonic electric toothbrush: Twice daily brushing
  Interventions: Device: Sonic electric toothbrush
- Manual toothbrush: Twice daily brushing
  Interventions: Device: Manual toothbrush

INTERVENTIONS:
Device: Oscillating-rotating electric toothbrush — Oscillating-rotating electric toothbrush used twice daily
  Groups: Oscillating-Rotating electric toothbrush
Device: Sonic electric toothbrush — Sonic electric toothbrush used twice daily
  Groups: Sonic electric toothbrush
Device: Manual toothbrush — Manual toothbrush used twice daily
  Groups: Manual toothbrush

SUMMARY:
The aim of this analysis was to compare gingivitis- and plaque-reduction efficacy from randomized controlled trials (RCTs) up to six months long evaluating oscillating-rotating, sonic, and manual toothbrushes

ELIGIBILITY:
Subjects were excluded from this study for the following reasons;

* pregnancy,
* rampant caries,
* severe periodontitis,
* at discretionary of the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This meta-analysis includes healthy adult male and females.
Sampling Method: Probability Sample
Enrollment: 2929 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Number of Bleeding Sites | Up to 6 months (26 weeks)
  Change from baseline as measured on number of bleeding sites ( via gingival bleeding index, Loe Silness index, Gingival Bleeding Index (GBI), Papillary bleeding index or Mazza gingival index).
Dental Plaque Scores | Up to 6 months (26 weeks)
  Change from baseline as measured by mean plaque score reduction from baseline (via Turesky's Modification of Quigley-Hein index, or Rustogi Modified Navy Plaque Index).

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Study Locations, Cincinnati, Ohio, United States